CLINICAL TRIAL: NCT03874689
Title: Establishment and Application of a Taenia Solium Experimental Pig Infection Model and Investigation of Environmental Factors Associated With Transmission of T. Solium in Endemic Villages of Eastern and Southern Provinces of Zambia
Brief Title: Investigation of Environmental Factors Associated With Transmission of T. Solium in Endemic Villages of Zambia
Acronym: TEPIM
Status: Completed | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: TEPIM
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Neurocysticercosis; Taeniosis
Keywords: Neurocysticercosis
MeSH Terms: conditions — Neurocysticercosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood and stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to determine the prevalence of taeniosis and (neuro)cysticercosis in two districts in the southern (Gwembe) and eastern province (Chipata) of Zambia.

DETAILED DESCRIPTION:
The true prevalence of Neurocyticercosis in Zambia is not well known. Only one study which was a pilot study done in Katete district of eastern province demonstrated the prevalence of NCC among people with epilepsy. There is need to provide an accurate estimate of the prevalence of NCC among people with cysticercosis in Zambia as well as understand the clinical manifestations of the disease in humans. Data on the full range of clinical characteristics of NCC is essential to accurately estimate the burden of the disease in the community.

The epidemiology work package within the human health sector will create awareness of the size of the problem by delivering scientifically generated prevalence data on TSCT and NCC in various population groups (adults, children, and those living with epilepsy) in two provinces of Zambia. This will form an essential prerequisite for the development of public health policy guidelines for the control/elimination of TSCT/NCC in the country.

Further, environmental factors that could play a role in the transmission and maintenance of T. solium eggs will be studied. This will provide essential data in understanding the epidemiology of the parasite in endemic regions.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to participate in all aspects of the study, including providing blood and stool samples, participating in a questionnaire survey and group discussions, and taking oral anthelmintic tablets
* Willing and able to provide informed consent (signature or thumbprint with impartial witness; assent for minors with parental consent).
* Living in, attending school in, or regularly visiting the bore holes present in, the study communities.
* Aged 10 years or older

Exclusion Criteria:

* Unwilling or unable to participate in some or all aspects of the study, including providing blood and stool samples, participating in a questionnaire survey and group discussions, or taking oral anthelmintic tablets.
* Unwilling or unable to provide written (signature or thumbprint with impartial witness) informed consent (or assent for minors).
* Living outside of, and not regularly visiting, or attending school in, the study communities.
* Children aged less than 10 years.
* Seriously ill individuals (people unable to engage in the normal activities of daily living without assistance because of their illnesses).

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study participants will be sampled from villages of two districts in Sambia (Gwembe and Chipata). Villages of these districts will be selected at random and all people from these villages will be invited to take part in the study. No selection apart from the exclusion criteria will take place.
Sampling Method: Probability Sample
Enrollment: 2921 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of T. solium cysticercosis | Assessment through blood sampling at baseline
  Prevalence of human T. solium cysticercosis
Prevalence of neurocysticercosis | Assessment at CT scanning at baseline
  Prevalence of human neurocysticercosis among people with positive serology for T. solium cysticercosis
Prevalence of taeniosis | Assessment through stool sampling at baseline
  Prevalence of human T. solium taeniosis

SECONDARY OUTCOMES:
Prevalence of intestinal helminth infection | Assessment through stool sampling at baseline
  Prevalence of intestinal helminth infection

CONTACTS AND LOCATIONS:
Overall Officials: Chummy S. Sikasunge, PhD, Principal Investigator — University of Zambia
Locations (1):
- University of Zambia, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zulu G, Sikasunge CS, Welte TM, Simuunza MC, Stelzle D, Schmidt V, Hachangu A, Mutale W, Masuku M, Chembensofu M, da Costa CP, Mwape KE, Winkler AS, Phiri IK. Epidemiology of intestinal helminthiasis with an emphasis on taeniasis in Chipata district of the Eastern province of Zambia. PLoS Negl Trop Dis. 2023 Nov 20;17(11):e0011561. doi: 10.1371/journal.pntd.0011561. eCollection 2023 Nov. PMID 37983246
- See also: Epidemiology of intestinal helminthiasis with an emphasis on taeniasis in Chipata district of the Eastern province of Zambia — https://journals.plos.org/plosntds/article?id=10.1371/journal.pntd.0011561